CLINICAL TRIAL: NCT01365013
Title: Effectiveness of the Translation of a Type 2 Diabetes Primary Prevention Program in Routine Context of Primary Heath Care
Brief Title: Evaluation of the Translation of the DE-PLAN Program for the Primary Prevention of Type 2 Diabetes in Routine Primary Care
Acronym: DE-PLAN E
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Carmen Silvestre Busto, Nurse, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010111039
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Prediabetic State
Keywords: Lifestyle; Prediabetic State; Patient Education; Primary Health Care
MeSH Terms: conditions — Prediabetic State | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: DE-PLAN
- control group (Active Comparator)
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: DE-PLAN — structured group or individual educational sessions (4 to 5) on diet and physical activity, plus ongoing reminder contacts (e-mails, sms, etc) during 1 year
  Arms: Lifestyle counseling
Behavioral: Control group — Standard advice for lifestyle change
  Arms: control group

SUMMARY:
The purpose of this study is to evaluate the feasibility and effectiveness of the DE-PLAN Euskadi program for the primary prevention of type-II diabetes in high-risk population seen in primary care centers (Osakidetza-Basque Health Service) in which such intervention is implemented, compared to usual care control centers.

DETAILED DESCRIPTION:
Objective: To evaluate the feasibility and effectiveness of the DE-PLANЄ program for the primary prevention of type-II diabetes in high-risk population seen in primary care centers (Osakidetza) in which such intervention is implemented, compared to usual care control centers.

DESIGN AND METHODS: A phase IV cluster randomized prospective clinical trial, conducted in 14 primary care centers from Osakidetza, which will be randomly assigned to intervention or control group, that will collect a sample of 2534 followed for two years, aged 45 to 70 years without diabetes but with high risk of developing it (FINDRISC scale> 14), identified by a screening system. Nurses in intervention centers (GI) will implement DEPLANЄ for 12 months, a structured educational intervention on healthy lifestyles (diet and physical activity), while patients of the control centers will receive standard care for the prevention and treatment of type-II diabetes.

ANALYSIS: The feasibility will be reported as the reach, adoption and implementation of the program. The attributable effectiveness of the program will be determined by comparing the changes in the incidence and risk of developing diabetes in healthy habits quality of life, observed in patients exposed to DE-PLANЄ intervention and of patients from control centers. The incremental cost-utility of DE-PLANЄ program will be also analysed.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 70 years old
* high risk of developing type-II diabetes (Findrisc scale > 14 points)

Exclusion Criteria:

* Disorders of the cardiovascular system
* Transplant recipients
* Renal or hepatic failure
* Severe chronic obstructive pulmonary disease
* Severe mental disorders
* Chronic and acute severe infections
* Metabolic uncontrolled disorders
* Restrictive pathology of muscles, bones and joints
* Complicated pregnancy
* Contact difficulties

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1113 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Adoption of healthy lifestyles | 12 months
  Change in the adoption of minimum recommended levels of physical activity and fruit and vegetable consumption
Incidence of Diabetes | 24 months
  Effectiveness of the program in the reduction of the Incidence of Diabetes

SECONDARY OUTCOMES:
Reach of the program | 24 months
  Percentage of eligible participants exposed to the program
Implementation of the program | 24 months
  Extent in which the intervention components have been delivered as intended (intervention protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Silvestre, Principal Investigator — Basque Health Service; Alvaro Sanchez, Principal Investigator — Basque Health Service
Locations (1):
- Primary Care Research Unit of Bizkaia, Bilbao, Spain

REFERENCES:
- [Derived] Sanchez A, Silvestre C, Campo N, Grandes G; PreDE research group. Type-2 diabetes primary prevention program implemented in routine primary care: a process evaluation study. Trials. 2016 May 20;17(1):254. doi: 10.1186/s13063-016-1379-0. PMID 27206733
- [Derived] Sanchez A, Silvestre C, Sauto R, Martinez C, Grandes G; PreDE research group. Feasibility and effectiveness of the implementation of a primary prevention programme for type 2 diabetes in routine primary care practice: a phase IV cluster randomised clinical trial. BMC Fam Pract. 2012 Nov 16;13:109. doi: 10.1186/1471-2296-13-109. PMID 23158830